CLINICAL TRIAL: NCT06924736
Title: Evaluate the Safety and Effectiveness of the Intravascular Shock Wave Treatment Device and the Disposable Coronary Intravascular Shock Wave Catheter Compared With the Non-compliant Balloon Catheter in the Treatment of In-stent Restenosis of the Coronary Artery
Brief Title: SONICURE（SONICracker for the Treatment of UndeRExpansion）
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Bluesail Boyuan Medical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LFBY-202503
Record Dates: First submitted 2025-03-17; First posted 2025-04-11 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-03

CONDITIONS: Coronary Artery Disease
Keywords: SONICURE
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intravascular Shockwave Therapy Device / Disposable Coronary Shockwave Catheter (Experimental): Intravascular Shockwave Therapy Device / Disposable Coronary Shockwave Catheter (Shanghai Lanfan Boyuan Medical Technology Co., Ltd.)
  Interventions: Device: Intravascular Shockwave Therapy Device / Disposable Coronary Shockwave Catheter
- non-compliant balloon dilatation catheter (Active Comparator): Randomized to the control group using a non-compliant balloon dilatation catheter (Shandong Jiwei Medical Products Co., Ltd.) to treat the lesion
  Interventions: Device: Non - compliant balloon dilatation catheter

INTERVENTIONS:
Device: Intravascular Shockwave Therapy Device / Disposable Coronary Shockwave Catheter — Randomly assign subjects to the experimental group to treat the lesions with an intravascular shockwave therapy device/disposable coronary artery shockwave catheter.
  Arms: Intravascular Shockwave Therapy Device / Disposable Coronary Shockwave Catheter
Device: Non - compliant balloon dilatation catheter — Randomly assign subjects to the control group to treat the lesions with a non - compliant balloon catheter.
  Arms: non-compliant balloon dilatation catheter

SUMMARY:
The first-phase study is a prospective, single-group observational study. It plans to recruit patients with in-stent restenosis caused by poor stent expansion in the coronary artery. The intravascular shock wave treatment device and the disposable coronary intravascular shock wave catheter produced by Shanghai Lifan Boyuan Medical Technology Co., Ltd. will be used for treatment. This is a clinical trial to verify the feasibility, preliminary safety and effectiveness of treating in-stent restenosis caused by poor stent expansion in the coronary artery.

The second-phase study is a prospective, multicenter, randomized controlled clinical trial is planned to recruit patients with in - stent restenosis caused by poor coronary stent expansion. These patients will be treated with either the intravascular shock wave treatment device and the disposable coronary intravascular shock wave catheter produced by Shanghai Lifan Boyuan Medical Technology Co., Ltd., or a non - compliant balloon dilation catheter (Shandong JW Medical Products Co., Ltd., National Medical Device Registration No. 20213031019). The purpose is to verify the safety and effectiveness of the investigational medical devices in treating in - stent restenosis caused by poor coronary stent expansion.

DETAILED DESCRIPTION:
In the first phase, it will be carried out at Beijing Luhe Hospital, Capital Medical University. A total of 10 subjects are planned to be enrolled. After the subjects are included in the study, they will be treated with the intravascular shock wave treatment device and the disposable coronary intravascular shock wave catheter produced by Shanghai Lifan Boyuan Medical Technology Co., Ltd. Clinical follow-ups will be conducted before discharge and one month after the operation.

In the second phase, it will be carried out at multiple clinical trial institutions in China. A total of 200 subjects are planned to be enrolled. After randomization, all subjects will undergo surgical treatment using either the investigational device or the control device. Clinical follow - up will be conducted before discharge, 1 month after surgery, and 6 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 80 years old, either male or non - pregnant female.
* Suffering from heart diseases with clinical evidence of ischemia, such as Chronic Coronary Syndrome (CCS) or Acute Coronary Syndrome (ACS).
* The subject should be able to understand the purpose of the trial, voluntarily participate in it, and sign the informed consent form.
* During the baseline surgery, at most one target lesion can be treated.
* The target lesion and non - target lesion are not located in the same blood vessel.
* The reference vessel diameter of the target lesion is 2.25 - 4.0 mm (estimated visually).

Exclusion Criteria:

* Patients who have had any myocardial infarction within 1 week, or patients who have had a myocardial infarction more than 1 week ago but whose myocardial enzymes CK or CK-MB have not yet returned to normal.
* Patients with New York Heart Association (NYHA) class III or IV heart failure or those with severe valvular heart disease.
* Female patients who are planning to become pregnant (or are breastfeeding).
* Severe impairment of liver and kidney function, with transaminase levels more than 3 times the upper limit of the normal value, serum creatinine > 2.5 mg/dL (221 μmol/L), or chronic renal failure requiring long-term dialysis.
* Severe hypertension that cannot be controlled despite treatment (systolic blood pressure persistently > 180 mmHg or diastolic blood pressure persistently > 110 mmHg).
* Coagulation disorders, with a platelet count < 100×10⁹/L.
* Patients with cardiogenic shock.
* Patients who need to receive cytostatic agents or radiotherapy due to accompanying diseases.
* Patients known to be allergic to heparin, contrast agents, aspirin, clopidogrel, or anesthetics.
* Patients with a bleeding diathesis, or those with a history of cerebral hemorrhage, active peptic ulcer, or gastrointestinal bleeding within the past 6 months, for whom anticoagulant therapy or the use of anticoagulant drugs will be restricted or prohibited.
* Patients with a life expectancy of less than 6 months or those with potential factors that may cause difficulties in clinical follow-up.
* Patients who are currently participating in any other clinical trial. Patients who, for other reasons, are considered by the investigator to be unsuitable for inclusion.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-05-15 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Surgical success rate | during the hospitalization period (up to 7 days after the operation).
  The residual stenosis after the operation is ≤ 30%, and there is no occurrence of Major Adverse Cardiac Events (MACE) during the hospitalization period (up to 7 days after the operation).

SECONDARY OUTCOMES:
Device success rate | Immediately after the operation
  Security endpoint
The minimum stent area immediately after the operation（MSA） | Immediately after the operation
  Measured by Optical Coherence Tomography (OCT)
The minimum stent lumen diameter immediately after the operation（MLD） | Immediately after the operation
  Measured by Optical Coherence Tomography (OCT)
The incidence of Major Adverse Cardiovascular Events (MACE) | before discharge, one month after the operation
  Safety endpoint
The incidence of target lesion failure (TLF) | one month after the operation
  Safety endpoint
The incidence of serious adverse events | before discharge, one month after the operation
  Safety endpoint
The incidence of device defects | during the operation
  Safety endpoint
The incidence of serious angiographic complications | during the operation
  Safety endpoint

CONTACTS AND LOCATIONS:
Overall Officials: Guangyao Zhai, Principal Investigator — Beijing Luhe Hospital Affiliated to Capital Medical University
Locations (1):
- Beijing Luhe Hospital Affiliated to Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No